CLINICAL TRIAL: NCT02458443
Title: Cardiovascular Response to Isometric Resistance Training in People With Hypertension for Blood Pressure Management
Brief Title: Isometric Handgrip Exercise for Blood Pressure Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New England, Australia (Other)
Responsible Party: Principal Investigator, Deb Carlson, Sponsor-Investigator, University of New England, Australia
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: UNewEngland
Record Dates: First submitted 2015-05-21; First posted 2015-06-01 (Estimated); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- IHG 5% Un-medicated (Sham Comparator): Participants with high blood pressure (greater than 120/80) who are not medicated for blood pressure control will conduct isometric handgrip (IHG) exercise at 5% of their maximum voluntary contraction (MVC). Isometric resistance training will be conducted three times a week for 12 weeks, with participants conducting 4 x 2min IHG exercises at each session.
  Interventions: Other: Isometric resistance training
- IHG 5% BB (Sham Comparator): Participants with high blood pressure (greater than 120/80) who are currently taking beta blockers for blood pressure control will conduct isometric handgrip exercise at 5% of their maximum voluntary contraction (MVC). Isometric resistance training will be conducted three times a week for 12 weeks, with participants conducting 4 x 2min IHG exercises at each session.
  Interventions: Other: Isometric resistance training
- IHG 30% Un-medicated (Experimental): Participants with high blood pressure (greater than 120/80) who are not medicated for blood pressure control will conduct isometric handgrip exercise at 30% of their maximum voluntary contraction (MVC). Isometric resistance training will be conducted three times a week for 12 weeks, with participants conducting 4 x 2min IHG exercises at each session.
  Interventions: Other: Isometric resistance training
- IHG 30% BB (Experimental): Participants with high blood pressure (greater than 120/80) who are currently taking beta blockers for blood pressure control will conduct isometric handgrip exercise at 30% of their maximum voluntary contraction (MVC). Isometric resistance training will be conducted three times a week for 12 weeks, with participants conducting 4 x 2min IHG exercises at each session.
  Interventions: Other: Isometric resistance training

INTERVENTIONS:
Other: Isometric resistance training — Isometric handgrip exercise using a hand dynamometer

SUMMARY:
Recent meta-analyses suggest isometric resistance training (IRT) may be superior to aerobic exercise for lowering blood pressure. The investigators intend to conduct the largest, longest, prospective, double-blind randomized controlled trial using isometric resistance training to reduce blood pressure to reduce hypertension.

DETAILED DESCRIPTION:
We are looking to assess the effect of isometric exercise on ambulatory blood pressure in participants aged 40-70 years who are either pre- or mild hypertensive; either un-medicated or taking medication to control their blood pressure. Our secondary aims are to examine whether the size of blood pressure change is different in those people taking or not taking anti-hypertensive medication, to determine the anti-hypertensive mechanism to IRT, and to establish rate of de-training effects after participants have ceased IRT.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure above 120/80 currently not taking anti-hypertensive medications whose doctor has suggested would benefit from exercise; and
* people currently taking beta blockers for blood pressure management.

Exclusion Criteria:

* Younger than 30yrs and older than 70 yrs;
* unable to voluntary participate;
* unable to participate under doctor's recommendation;
* smokers;
* arthritis or carpal tunnel which may be aggravated with handgrip exercise;
* known cardiovascular disease (angina) and the following co-morbid conditions:

  * obesity,
  * insulin resistance,
  * depression,
  * mobility impairment,
  * sleep apnoea,
  * fatty liver disease or
  * renal disease

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in systolic and diastolic blood pressure | Change measures: baseline and 12 weeks

SECONDARY OUTCOMES:
Compare and contrast change in systolic and diastolic blood pressure of medicated and un-medicated participants | Baseline and 12 weeks
Detraining effects, changes in systolic and diastolic blood pressure after cessation of Isometric Resistance Training | 12 weeks and 24 weeks
  End of exercise protocol and 12 weeks after completion

CONTACTS AND LOCATIONS:
Overall Officials: Neil Smart, PhD, Principal Investigator — University of New England
Locations (1):
- UNE Exercise Physiology Lab, Armidale, New South Wales, Australia

REFERENCES:
- [Background] Carlson DJ, Dieberg G, Hess NC, Millar PJ, Smart NA. Isometric exercise training for blood pressure management: a systematic review and meta-analysis. Mayo Clin Proc. 2014 Mar;89(3):327-34. doi: 10.1016/j.mayocp.2013.10.030. PMID 24582191